CLINICAL TRIAL: NCT05070689
Title: Placenta Accreta Spectrum Disorders: A. Chohan Continuous Squeezing Suture (ACCSS) for Controlling Haemorrahge From Lower Uterine Segment at Caesarean Section
Brief Title: Placenta Accreta Spectrum Disorders: A. Chohan Continuous Squeezing Suture (ACCSS)
Acronym: ACCSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sharif Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMDC/SMRC/209-21
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-08

CONDITIONS: Placenta Accreta
Keywords: Peripartum Hystrectomy; Postpartum Haemorrhage
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): A. Chohan Continuous squeezing Suture (ACCSS): An obstetrical procedure using half circle 40mm round body polyglactin 910 suture # 1 (Vicryl plus by Ethicon ®) for control of haemorrhage from the lower segment, in patients with Placenta Accreta for the prevention of hysterectomy at caesarean section
  Interventions: Procedure: ACCSS

INTERVENTIONS:
Procedure: ACCSS — A. Chohan Continuous Squeezing Suture (ACCSS)

SUMMARY:
Placenta Accreta Spectrum (PAS) disorders are rising in incidence due to increased rate of repeat caesarean sections. Peripartum hysterectomy remains the only definitive treatment of massive postpartum haemorrhage related to this condition. Researchers have described conservative treatments in the form of pelvic devascularization under radiological control, myometrial resection with placenta in situ, and various suturing techniques some involving inversion of cervix. Variable success rates are described, but search continues for a simple, safe and effective treatment. The objective of this study is to assess the simplicity, safety and efficacy of A. Chohan Continuous Squeezing Suture (ACCSS) in the management of PAS.

DETAILED DESCRIPTION:
Placenta accreta spectrum has opened up a new era in the history of PPH, as forcible separation of adherent placenta leads to massive bleeding from placental bed . Peripartum hysterectomy has emerged as gold standard treatment for this variety of PPH (3 folds rise over uterine atony) with its overall morbidity of 40-50%, and mortality of 7-10% in case of placenta percreta . The fear of placental bed bleeding has led to the development of conservative management like "leaving the placenta in situ approach" with its wide range of mild to severe, and serious morbidities . The conservative surgical techniques (The triple P procedure, one step conservative surgery approach) have also used the concept of non-separation of placenta and have instead adopted resection of myometrium with placenta in situ . These surgeries involve devascularisation of deep pelvic / major abdominal vessels and ligation of complex arterial anastomosis making the procedure technically difficult. Moreover, the devascularisation is done under extensive and expensive interventional radiological equipment which places the procedures out of reach for the routine setups particularly in the under developed countries. Another conservative surgical technique (stepwise surgical approach) , which described separation of placenta also mainly relied upon devascularisation of pelvic organs by bilateral ligation of anterior branch of internal iliac artery rather than elaborating the details of technique of controlling haemorrhage at the actual bleeding site.

Rationale of ACCSS ACCSS is a novel suturing technique addresses the management of placenta praevia and PAS following the orthodox approach of separation of placenta, taking the challenge of controlling massive haemorrhage. The rational of ACCSS is; i. Placental bed is the ultimate area of concern in women with placenta praevia and PAS, and it generally spreads over the whole inner surface of lower uterine segment, but the placental attachment and bleeding area upon its separation does not extend onto the internal os and into the vagina.

ii. Lower uterine segment is thin, flexible, squeezable and holds the suture well.

iii. Internal cervical os is a fixed structure, and has a ring with sufficient strength to function as anchor to the suture.

iv. Taking half thickness of internal cervical os into suture does not alter the anatomy and uterine drainage remains unaffected.

v. Deep pelvic devascularization by ligation or balloon tamponade occlusion (under radiological control) of deep pelvic vessels was not the part of ACCSS procedure. Bilateral uterine artery ligation was added to it because occlusion of the uterine artery or its branches is useful procedure to stop upper uterine bleeding , it does not appear to affect fertility or obstetric outcome and vascular occlusion is only temporary, as recanalization soon ensures normal uterine circulation . The haemostatic effect of ACCSS is therefore independent and does not rely upon supportive measures.

SURGICAL PROCEDURE The caesarean sections in this study will be performed between 37 and 38 weeks of gestation on all patients. Haematology department will be placed on alert with availability of 4 units of cross matched fresh blood and fresh frozen plasma. All surgeries will be performed by principal investigators (Prof Dr. Arshad Chohan & Prof. Dr. Fauzia). A multidisciplinary team comprising of experienced obstetricians, anaesthetist, and paediatrician will be involved during the procedure. Prophylactic antibiotic (ceftriaxone 1gm intravenously) will be administered to all patients before surgery.

At caesarean section Pfannenstiel incision will be used for all patients. After opening the abdomen, a clinical assessment about the depth of invasion of the placenta will be made to exclude the involvement of bladder and other pelvic organs. The features noted at this assessment will be abnormal placental bulge and hypervascularity on uterine serosal surface, and placental invasion into the urinary bladder and/or other pelvic organs. Prior to uterine incision placental site will be gently reconfirmed with the examining hand to ascertain an easy fetal access and to avoid cutting of placenta particularly in case of anterior dominant placenta. A transverse incision will be given in the lower uterine segment (LUS) above the insertion of placenta and the baby will be delivered. At delivery of baby10 iu of oxytocin will be given intravenously, followed by 40 iu in 500 ml of normal saline at the rate of 125ml/hour for first 24 hours as per hospital policy for caesarean section for PAS. The uterus will be exteriorized without making any efforts to remove the placenta. The bleeding edges of the uterine incision will be held with Green-Armitage forceps to minimize bleeding. The visceral peritoneum will be displaced downwards with sharp and blunt dissection to allow suturing on the inner side of the LUS. Bladder will be dissected away only if found adherent with the lower uterine segment from previous caesarean sections. Uterine arteries will be ligated on both sides and any blood vessels on the way will be secured. The placenta will then be removed to as close to complete as possible. The lower uterine segment will be packed with sponge to arrest haemorrhage temporarily while preparing for the suture.

ACCSS Application The packing will be removed and the ring of internal os will be identified with the index and middle finger of one hand and held with Babcock forceps with the other hand. On the exposed inner surface of the LUS, suturing will be started from the left corner of uterine incision, using half circle 40mm round body polyglactin 910 suture # 1 (vicryl plus by Ethicon ®) taking multiple half cm bites through half-thickness of the tissue at half cm intervals to reach the outer half of ring of internal os. The suture will then tied and first knot secured causing squeezing of uterine tissue. From here onwards similar sutures will be placed continuously at 1 cm distance till the right corner will be reached, where the second knot will be secured. During suturing the patency of the internal os will be ensured. The continued pull on the suture is expected to cause squeezing of the LUS and arrest bleeding from all sinuses present at the placental site . A similar suture will be applied on the posterior uterine wall in case of bleeding from posterior uterine wall. The suture will be started from the outer half of the posterior lip of the ring of the internal os and going up to the highest bleeding point on the posterior wall of the uterus, continuing from the left to right end of the uterine incision . Any leftover bleeding points will be secured with separate sutures to ensure complete haemostasis. The uterine incision will be closed in two layers as done in a routine lower segment caesarean section. Any additional medical or surgical therapy instituted will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. The women at 32 weeks' gestation with central (anterior dominant, posterior) placenta praevia.
2. The women with Placenta Accreta Spectrum disorders having myometrial invasion limited to the uterine serosa (Grade 1, 2, and 3a) without involvement of urinary bladder and other pelvic organs.
3. The women wishing to conserve the uterus at the time of caesarean section.

Exclusion Criteria:

1. The patients with placenta accreta spectrum disorder with bladder and other organs involvement (Grade 3b, 3c) diagnosed prenatally and during caesarean section.
2. The patients with laterally situated right and left placentae.
3. The recruited patients who required emergency caesarean section.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-14 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Peripartum Hysterectomy | 24 hours
  Absolute number of peripartum hysterectomies within the study group

SECONDARY OUTCOMES:
Application time of suture in minutes | within 20 minutes
  Application time of suture plus time to complete haemostasis in minutes
Estimated blood loss | First 24 hours
  Estimate of blood loss in milliliters (ml) intraoperatively and within first 24 hours
Number of units of blood transfusions | First 24 hours
  Number of blood transfusions intraoperatively and within first 24 hours
Intensive care unit admissions | 7 days
  Number of days of admission in Intensive care unit
Duration of stay in hospital | 7 days
  Duration of stay in hospital in days
Urinary tract trauma and its complication | 6 weeks
  Bladder trauma/ vesicovaginal fistula
Uterine complications | 6 weeks
  Uterine necrosis/abscess formation
Secondary postpartum hemorrhage | 6 weeks
  Abnormal uterine bleeding within 6 weeks
Maternal mortality | 6 weeks
  Number of mothers dying in relation to cesarean section within 6 completed weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Arshad Chohan, FRCOG, Principal Investigator — Sharif Medical And Dental College
Locations (1):
- Sharif Medical and Dental college, Lahore, Pakistan/Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ngwenya S. Postpartum hemorrhage: incidence, risk factors, and outcomes in a low-resource setting. Int J Womens Health. 2016 Nov 2;8:647-650. doi: 10.2147/IJWH.S119232. eCollection 2016. PMID 27843354
- [Result] Jauniaux E, Gronbeck L, Bunce C, Langhoff-Roos J, Collins SL. Epidemiology of placenta previa accreta: a systematic review and meta-analysis. BMJ Open. 2019 Nov 12;9(11):e031193. doi: 10.1136/bmjopen-2019-031193. PMID 31722942
- [Result] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Result] Huque S, Roberts I, Fawole B, Chaudhri R, Arulkumaran S, Shakur-Still H. Risk factors for peripartum hysterectomy among women with postpartum haemorrhage: analysis of data from the WOMAN trial. BMC Pregnancy Childbirth. 2018 May 29;18(1):186. doi: 10.1186/s12884-018-1829-7. PMID 29843627
- [Result] Palacios-Jaraquemada JM, Fiorillo A, Hamer J, Martinez M, Bruno C. Placenta accreta spectrum: a hysterectomy can be prevented in almost 80% of cases using a resective-reconstructive technique. J Matern Fetal Neonatal Med. 2022 Jan;35(2):275-282. doi: 10.1080/14767058.2020.1716715. Epub 2020 Jan 26. PMID 31984808